CLINICAL TRIAL: NCT00898040
Title: Proposal for Combining ECOG Myeloma Trial SNP Data
Brief Title: Study of DNA Samples From Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Other Study IDs: CDR0000495284; ECOG-E3L06T1
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; refractory multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective

INTERVENTIONS:
Genetic: polymorphism analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that may occur in DNA and identify biomarkers related to cancer.

PURPOSE: This laboratory study is looking at DNA samples from patients with multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether there is an increased frequency of 1 or more polymorphic alleles that are associated with clinical endpoints using custom myeloma single nucleotide polymorphism (SNP) chip analysis of banked DNA samples from patients with multiple myeloma.
* Determine SNPs associated with toxicities caused, not by variations in tumor cell genetics, but by individual genetic variations affecting drug activation, distribution, metabolism, and export (ADME).
* Determine SNPs associated with response, influenced by the same ADME.
* Determine SNPs associated with bone disease (as a variable) among patients with multiple myeloma.
* Determine SNPs associated with epidemiology (i.e., risk factors for the development of multiple myeloma).

OUTLINE: This is a retrospective, multicenter study.

Banked DNA samples are analyzed using a custom single nucleotide polymorphism (SNP) chip to assess approximately 3,590 SNPs from 1,061 genes that are associated with myeloma growth and response.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma
* DNA samples banked from other ECOG studies (and other clinical trial groups [e.g., SWOG and MRC])

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-07-06 (Actual); Primary Completion 2007-01-01 (Actual); Study Completion 2007-01-01 (Actual)

PRIMARY OUTCOMES:
Increased frequency of ≥1 polymorphic alleles associated with clinical endpoints using custom myeloma SNP chip analysis of banked DNA samples from patients with multiple myeloma | 1 month
SNPs associated with toxicities caused by individual genetic variations affecting drug activation, distribution, metabolism, and export (ADME) | 1 month
SNPs associated with response | 1 month
SNPs associated with bone disease | 1 month
SNPs associated with epidemiology (i.e., risk factors for the development of multiple myeloma) | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Brian Van Ness, Study Chair — Masonic Cancer Center, University of Minnesota